CLINICAL TRIAL: NCT00813423
Title: Autophagic Modulation With Anti-angiogenic Therapy in Patients With Advanced Malignancies: A Phase I Trial of Sunitinib and Hydroxychloroquine
Brief Title: Sunitinib Malate and Hydroxychloroquine in Treating Patients With Advanced Solid Tumors That Have Not Responded to Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03112; NCI-2012-03112 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CTEP #8342; 050909 (Other: Rutgers Cancer Institute of New Jersey); 8342 (Other: CTEP); P30CA072720 (NIH); U01CA132194 (NIH)
Record Dates: First submitted 2008-12-20; First posted 2008-12-23 (Estimated); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Adult Solid Neoplasm
MeSH Terms: interventions — Hydroxychloroquine; Sunitinib

ARMS (1):
- Treatment (sunitinib malate, hydroxychloroquine) (Experimental): Patients receive sunitinib malate PO QD on days 1-28 and hydroxychloroquine PO QD or BID on days 1-42 (beginning day 4 of course 1). Treatment repeats every 42 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Hydroxychloroquine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sunitinib Malate

INTERVENTIONS:
Drug: Hydroxychloroquine — Given PO
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Sunitinib Malate — Given PO
  Other Names: SU011248; SU11248; sunitinib; Sutent

SUMMARY:
This phase I trial studies the side effects and best dose of sunitinib malate when given together with hydroxychloroquine in treating patients with advanced solid tumors that have not responded to chemotherapy. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Hydroxychloroquine may help sunitinib malate work better in treating solid tumors. Giving sunitinib malate together with hydroxychloroquine may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of the combination of sunitinib (sunitinib malate) (Sutent), an oral tyrosine kinase inhibitor with antiangiogenic activity that inhibits vascular endothelial growth factor receptor 2 (VEGFR2), stem cell factor receptor (c-kit) and platelet derived growth factor receptor (PDGFR), in combination with hydroxychloroquine (HCQ), an inhibitor of autophagy, in patients with advanced solid tumors that are refractory to standard chemotherapy.

SECONDARY OBJECTIVES:

I. Evaluating blocks of tissue from pre-treatment diagnostic biopsies and tissue from biopsies taken during therapy, when available from enrolled patients, for expression of markers beclin1, light chain 3 (LC3), sequestosome 1 (p62) and hypoxia up-regulated 1 (GRp170) as indicators of autophagy potential.

II. Evaluating pre- and post- treatment peripheral blood mononuclear cells (PBMC) and tumor tissue, when available, for the presence of autophagosomes by electron microscopy (EM) as indication of flux through the autophagy pathway.

III. Evaluating pre- and post- treatment PBMC for changes in the expression of LC3, p62 and GRp170 with the use of single agent sunitinib and the use of the combination of sunitinib with hydroxychloroquine.

IV. Evaluating circulating tumor cells (CTCs) pre- and post- treatment with single agent sunitinib and sunitinib + HCQ, and characterize these for markers of autophagy. (exploratory) V. To determine whether the steady-state plasma concentration of HCQ correlates with inhibition of autophagy and whether a pharmacokinetic interaction exists between sunitinib and HCQ.

VI. To examine, when available, post treatment tumor biopsies for vascular markers to detect decreased vascular proliferation by staining cluster of differentiation 31 (CD31), vascular endothelial growth factor (VEGF), thrombospondin-1, and cluster of differentiation 105 (CD105) staining to monitor micro vessel density.

OUTLINE: This is a dose-escalation study of hydroxychloroquine.

Patients receive sunitinib malate orally (PO) once daily (QD) on days 1-28 and hydroxychloroquine PO once daily (QD) or twice daily (BID) on days 1-42 (beginning day 4 of course 1). Treatment repeats every 42 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically proven advanced cancer
* Patients must have undergone treatment with at least one regimen of standard therapy, either cytotoxic chemotherapy, an oral targeted agent or immunotherapy, or have a form of cancer for which no standard therapy exists, or are not eligible for or decline standard therapy; patients who have received prior therapy with sunitinib will be allowed; patients with prostate cancer may continue on hormonal therapy if they are currently receiving it
* Patients must have measurable or evaluable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Life expectancy > 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Serum calcium =< 12.0 mg/dL
* Total serum bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/ananine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal, unless the patient has liver metastases, in which case both AST and ALT must be =<5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Thyroid-stimulating hormone (TSH) within normal institutional limits is required for eligibility; free T3 and free T4 values will also be obtained for baseline values should repeat parameters be required later in the course of treatment, however these values will not be used to determine eligibility
* Creatine phosphokinase (CPK) within normal institutional limits
* The following groups of patients are eligible provided they have New York Heart Association class II (NYHA) cardiac function on baseline echocardiogram (ECHO)/multi gated acquisition scan (MUGA):

  * Those with a history of class II heart failure who are asymptomatic on treatment
  * Those with prior anthracycline exposure
  * Those who have received central thoracic radiation that included the heart in the radiotherapy port
* Patients who require use of therapeutic doses of Coumadin-derivative anticoagulants such as warfarin are excluded, although doses of up to 2 mg daily are permitted for prophylaxis of thrombosis; note: low molecular weight heparin is permitted provided the patient's prothrombin time (PT) international normalized ratio (INR) is =< 1.5
* Ejection fraction measured within institutional limits of normal by MUGA scan
* Patients with known brain metastases should be excluded because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Women must: Have a negative serum or urine pregnancy test within 7 days prior to study entry if she is a woman of child-bearing potential (WOCBP), OR

  * Be at least one year post-menopausal, OR
  * Be surgically sterile
* Patients of childbearing or child fathering potential must be willing to use an acceptable method of birth control prior to study entry and for the duration of the study; acceptable methods of contraception include hormonal, barrier methods, intrauterine device, tubal ligation/vasectomy or abstinence; women should not breast feed while on treatment with sunitinib and HCQ
* Patients must not have a history of any condition (social or medical) that, in the opinion of the investigator, might interfere with the patient's ability to comply with the protocol or pose additional or unacceptable risk to the patient
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain sunitinib tablets are excluded
* Approval for HCQ treatment by an eye doctor, based on a screening eye exam; examples of disqualifying baseline conditions include macular degeneration and other retinal disease, see exclusion criteria
* Patients must be able to understand and sign informed consent

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy or biologic agents within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; at least 4 weeks must have elapsed since any major surgery
* Patients on treatment for rheumatoid arthritis or systemic lupus erythematosus
* Patients receiving any disease-modifying anti-rheumatic drug (DMARD)
* Active clinically significant infection requiring antibiotics, antivirals or antifungals; these medications may be allowed for instances of prophylaxis or treatment felt to not be clinically significant at the discretion of the principal investigator
* Patients with poorly controlled hypertension (systolic blood pressure of 140 mmHg or higher or diastolic blood pressure of 90 mmHg or higher) are ineligible
* Patients with a pre-existing thyroid abnormality who are unable to maintain thyroid function in the normal range with medication are ineligible
* Diagnosis or history of central nervous system (CNS) disease (i.e. primary brain tumor, malignant seizures, untreated CNS metastases or carcinomatous meningitis or CNS metastases)
* Patient must not have ongoing ventricular cardiac dysrhythmias of grade = 2 as described by the Cancer Therapy Evaluation Program (CTEP) Active Version of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE); patients with a history of serious ventricular arrhythmia (ventricular tachycardia [VT] or ventricular fibrillation [VF] > 3 beats in a row) are also excluded; additionally, patients with ongoing atrial fibrillation are not eligible
* Corrected QT (QTc) interval >= 500 msec on baseline electrocardiogram (EKG)
* Any of the following within 6 months prior to first dose of treatment: myocardial infarction, symptomatic coronary artery disease (severe or unstable angina), artery bypass graft, uncontrolled arrhythmias, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolus
* Patients with known human immunodeficiency virus (HIV) are excluded due to possibility of unknown side effects on the immune system by these agents; the potential impact of pharmacokinetic interactions of retroviral therapy with sunitinib is unknown; appropriate studies may be undertaken in patients with HIV and those receiving combination anti-retroviral therapy in the future
* Because sunitinib is metabolized primarily by the cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) liver enzyme, the eligibility of patients taking medications that are potent inducers or inhibitors of that enzyme will be determined following a review of their case by the principal investigator; every effort should be made to switch patients taking such agents or substances to other medications
* Must not have psoriasis or porphyria
* Must not have known hypersensitivity to 4-aminoquinoline compound
* Must not have retinal or visual field changes from prior 4-aminoquinoline compound use
* Must not have known glucose-6-phosphate dehydrogenase (G-6PD) deficiency
* Patients must not have any known gastrointestinal (GI) pathology that would interfere with drug bioavailability
* Patients must not have known prior hypersensitivity to sunitinib or hydroxychloroquine or any of their components
* Must not be taking hydroxychloroquine for treatment or prophylaxis of malaria
* Patients must not have a clinically significant bleeding or clotting disorder
* Patients requiring medication with aurothioglucose (contraindicated with concurrent administration of antimalarials)
* History of gastrointestinal perforation, or intra-abdominal abscess within the previous 28 days
* Serious, non-healing infection, bone fracture or nonhealing ulcer or wound
* Current treatment on another clinical trial; participation in non-therapeutic clinical trials is permissible
* Patients with nephrotic syndrome
* Cataracts that would interfere with required funduscopic examinations, or severe baseline visual impairment including macular degeneration, retinopathy or visual field changes, or having only one functional eye; all patients must undergo a screening eye exam prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02-19 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
MTD of sunitinib malate, as assessed by the NCI CTCAE version 4.0 (v4.0) | 28 days
Response rate using the international criteria RECIST | Up to 2 years
  Reported with 95% confidence interval.

SECONDARY OUTCOMES:
Survival | Up to 2 years
  Analyzed using Kaplan-Meier product limit method.
Percent changes of the marker expressions, beclin1, LC3, p62 and GRp170, as indicators of autophagy potential in tissue | Up to 96 hours post-dose (course 2)
  Mean or median changes estimated by t-test or Wilcoxon signed rank test. Multiple test adjustment will be considered to control the overall type-I error rate.
Mean number of autophagic vesicles per cell (mAV/cell) by electron microscopy (EM) as indication of flux through the autophagy pathway for non-apoptotic cells | Up to 96 hours post-dose (course 2)
  Perform using a (pre-post samples) paired t-test.
Steady-state plasma concentration of hydroxychloroquine (HCQ) | Up to 96 hours post-dose (course 2)
  The correlation between the steady-state plasma concentration of HCQ and of autophagy inhibition and pharmacokinetic (PK) interaction will be assessed by regression analyses with treatment (sunitinib malate and +HCQ) as a stratification covariate in the model.
Autophagy inhibition and PK interaction | Up to 96 hours post-dose (course 2)
  The correlation between the steady-state plasma concentration of HCQ and of autophagy inhibition and PK interaction will be assessed by regression analyses with treatment (sunitinib malate and +HCQ) as a stratification covariate in the model.
Percent changes of the vascular marker levels of CD31, VEGF, thrombospondin-1, and CD105 for detection of decreased vascular proliferation | Up to 96 hours post-dose (course 2)
  Mean or median changes examined by t-test or Wilcoxon signed rank test. Multiple test adjustment will be considered to control the overall type-I error rate.

CONTACTS AND LOCATIONS:
Overall Officials: Janice M Mehnert, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey